CLINICAL TRIAL: NCT06705426
Title: Scapular Mobilization Versus Posterior Capsular Stretch in Frozen Shoulder
Brief Title: Scapular Mobilization Versus Capsular Stretch
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia Ahmed Abd Elmeged, Principal Investiator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005349
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-11

CONDITIONS: Frozen Shoulder
MeSH Terms: conditions — Bursitis | interventions — Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Scapular mobilization group A (Experimental): Scapular mobilization with addition anterior, posterior ,caudal glenohumeral mobilization, infrared therapy, ultrasound therapy, pendulum exercises
  Interventions: Other: Scapular mobilization with addition anterior, posterior ,caudal glenohumeral mobilization, infrared therapy, ultrasound therapy, pendulum exercises
- Posterior capsular stretch group B (Experimental): Posterior capsular stretch with addition anterior, posterior ,caudal glenohumeral mobilization, infrared therapy, ultrasound therapy, pendulum exercises
  Interventions: Other: Posterior capsular stretch with addition anterior, posterior ,caudal glenohumeral mobilization, infrared therapy, ultrasound therapy, pendulum exercises

INTERVENTIONS:
Other: Scapular mobilization with addition anterior, posterior ,caudal glenohumeral mobilization, infrared therapy, ultrasound therapy, pendulum exercises — Scapular mobilization with addition anterior, posterior ,caudal glenohumeral mobilization, infrared therapy, ultrasound therapy, pendulum exercises
  Arms: Scapular mobilization group A
Other: Posterior capsular stretch with addition anterior, posterior ,caudal glenohumeral mobilization, infrared therapy, ultrasound therapy, pendulum exercises — Posterior capsular stretch with addition anterior, posterior ,caudal glenohumeral mobilization, infrared therapy, ultrasound therapy, pendulum exercises
  Arms: Posterior capsular stretch group B

SUMMARY:
The goal of this study is to compare the effect of scapular mobilization versus posterior capsular stretch on pain, function, range of motion, and posterior capsular tension in patient with frozen shoulder

DETAILED DESCRIPTION:
Frozen shoulder is a musculoskeletal condition that is commonly encountered in physical therapy practice. It is characterized by a painful, gradual loss of both active and passive glenohumeral motion resulting from progressive fibrosis and ultimate contracture of the glenohumeral joint capsule. Frozen shoulder affects about 2% of the general population, with a higher prevalence in people between their 40s and 60s. Frozen shoulder occurs more in diabetic patient.

The traditional principles of treatment of frozen shoulder are to relieve pain, maintain range of motion, and ultimately to restore function. The physiotherapy treatment of frozen shoulder consists of different modalities such as Transcutaneous Electrical Nerve Stimulation (TENS), Interferential Therapy (IFT), Ultrasound, Short Wave Diathermy (SWD) etc., and the physical therapy exercises such as stretching, Codman exercise can be used.

Scapular-mobility exercises, or scapular-mobilization (SM) techniques is widely used in the management of musculoskeletal disorders of the shoulder. Scapular mobilization can cause pain reduction with improvement in the shoulder range of motion. Scapular mobilization can reduce the disability in patients with shoulder dysfunction.

Posterior capsular stretch is applied along with mobilization which causes significant improvement in increasing range of motion and functional disability. Capsular stretching showed a more significant reduction in pain when compared to general exercises.

Therefore, what are the possible effect of scapular mobilization versus posterior capsular stretch in treating patients with frozen shoulder?

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged from 40-65 years old.
* Diabetic and non-diabetic patients' diagnosis of stage 3 frozen shoulder (frozen phase) by an orthopedist.
* The presence of pain and limited movement in the shoulder for at least 2 months.
* Passive joint movements are limited when compared with the normal side.
* Unilateral involvement.

Exclusion Criteria:

* Recent joint infection or surgery.
* History of shoulder subluxation, dislocation, or ligamentous injury.
* Shoulder arthroplasty.
* Shoulder and cervical pathology.
* Recent trauma.
* Neurological disorders with muscle weakness in the shoulder joint.
* Infection, pregnancy, carcinoma patients, severe cardiac or psychiatric conditions.
* Previous shoulder surgeries to the affected shoulder.
* Previous manipulations under anesthesia of the affected shoulder.
* Radiological evidence for glenohumeral joint arthritis.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Shoulder flexion range of motion to measure shoulder joint active range of motion (flexion) by bubble inclinometer | pre-intervention, after 2 weeks of treatment and post treatment 4 weeks
Shoulder abduction range of motion to measure shoulder joint active range of motion (abduction) by bubble inclinometer | pre-intervention, after 2 weeks of treatment and post treatment 4 weeks
Shoulder internal rotation range of motion to measure shoulder joint active range of motion (internal rotation) by bubble inclinometer | pre-intervention, after 2 weeks of treatment and post treatment 4 weeks
Shoulder external rotation range of motion to measure shoulder joint active range of motion (external rotation) by bubble inclinometer | pre-intervention, after 2 weeks of treatment and post treatment 4 weeks
Shoulder pain and disability index to measure the shoulder pain the maximum possible score for the pain scale is 50 | pre-intervention, after 2 weeks of treatment and post treatment 4 weeks
Shoulder pain and disability index to measure the disability level the maximum possible score for the disability scale is 80 | pre-intervention, after 2 weeks of treatment and post treatment 4 weeks
poaterior capsular tension measurement by ruler | pre-intervention, after 2 weeks of treatment and post treatment 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karima A Hassan, Principal Investigator — Karima.abdelaty@pt.cu.edu.eg

REFERENCES:
- [Background] Ali SA, Khan M. Comparison for efficacy of general exercises with and without mobilization therapy for the management of adhesive capsulitis of shoulder - An interventional study. Pak J Med Sci. 2015 Nov-Dec;31(6):1372-6. doi: 10.12669/pjms.316.7909. PMID 26870099
- [Background] Duzgun I, Baltaci G, Atay OA. Manual therapy is an effective treatment for frozen shoulder in diabetics: an observational study. Eklem Hastalik Cerrahisi. 2012;23(2):94-9. PMID 22765488
- [Background] Duzgun I, Turgut E, Eraslan L, Elbasan B, Oskay D, Atay OA. Which method for frozen shoulder mobilization: manual posterior capsule stretching or scapular mobilization? J Musculoskelet Neuronal Interact. 2019 Sep 1;19(3):311-316. PMID 31475938
- [Background] Kurtais Gursel Y, Ulus Y, Bilgic A, Dincer G, van der Heijden GJ. Adding ultrasound in the management of soft tissue disorders of the shoulder: a randomized placebo-controlled trial. Phys Ther. 2004 Apr;84(4):336-43. PMID 15049727
- [Background] Klauser AS, Tagliafico A, Allen GM, Boutry N, Campbell R, Court-Payen M, Grainger A, Guerini H, McNally E, O'Connor PJ, Ostlere S, Petroons P, Reijnierse M, Sconfienza LM, Silvestri E, Wilson DJ, Martinoli C. Clinical indications for musculoskeletal ultrasound: a Delphi-based consensus paper of the European Society of Musculoskeletal Radiology. Eur Radiol. 2012 May;22(5):1140-8. doi: 10.1007/s00330-011-2356-3. Epub 2012 Mar 28. PMID 22453857
- [Background] Laudner KG, Sipes RC, Wilson JT. The acute effects of sleeper stretches on shoulder range of motion. J Athl Train. 2008 Jul-Aug;43(4):359-63. doi: 10.4085/1062-6050-43.4.359. PMID 18668168
- [Background] Leung MS, Cheing GL. Effects of deep and superficial heating in the management of frozen shoulder. J Rehabil Med. 2008 Feb;40(2):145-50. doi: 10.2340/16501977-0146. PMID 18509580
- [Background] Le HV, Lee SJ, Nazarian A, Rodriguez EK. Adhesive capsulitis of the shoulder: review of pathophysiology and current clinical treatments. Shoulder Elbow. 2017 Apr;9(2):75-84. doi: 10.1177/1758573216676786. Epub 2016 Nov 7. PMID 28405218
- [Background] Lewis J. Frozen shoulder contracture syndrome - Aetiology, diagnosis and management. Man Ther. 2015 Feb;20(1):2-9. doi: 10.1016/j.math.2014.07.006. Epub 2014 Jul 18. PMID 25107826
- [Background] McClure P, Balaicuis J, Heiland D, Broersma ME, Thorndike CK, Wood A. A randomized controlled comparison of stretching procedures for posterior shoulder tightness. J Orthop Sports Phys Ther. 2007 Mar;37(3):108-14. doi: 10.2519/jospt.2007.2337. PMID 17416125
- [Background] Paul A, Rajkumar JS, Peter S, Lambert L. Effectiveness of sustained stretching of the inferior capsule in the management of a frozen shoulder. Clin Orthop Relat Res. 2014 Jul;472(7):2262-8. doi: 10.1007/s11999-014-3581-2. Epub 2014 Mar 25. PMID 24664198
- [Background] Surenkok O, Aytar A, Baltaci G. Acute effects of scapular mobilization in shoulder dysfunction: a double-blind randomized placebo-controlled trial. J Sport Rehabil. 2009 Nov;18(4):493-501. doi: 10.1123/jsr.18.4.493. PMID 20108851
- [Background] Zuckerman JD, Rokito A. Frozen shoulder: a consensus definition. J Shoulder Elbow Surg. 2011 Mar;20(2):322-5. doi: 10.1016/j.jse.2010.07.008. Epub 2010 Nov 4. PMID 21051244